CLINICAL TRIAL: NCT05756946
Title: Guided Tissue Regeneration Combined With Periodontal Dressing: A Randomized Controlled Clinical Trial for the Treatment of Periodontal Defects
Brief Title: Guided Tissue Regeneration With a Periodontal Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Ta'a, Associate Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GTR
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Periodontal Dressings; Coe-Pak; Guided Tissue Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test group will receive GTR + periodontal dressing (Coe-pak)
  Interventions: Procedure: periodontal dressing (coe-pak); Procedure: Guided Tissue Regeneration
- Control group (Active Comparator): Control group will receive GTR only
  Interventions: Procedure: Guided Tissue Regeneration

INTERVENTIONS:
Procedure: periodontal dressing (coe-pak) — Guided tissue regeneration and periodontal dressing
  Arms: Test group
Procedure: Guided Tissue Regeneration — Regeneration of lost periodontal tissues
  Other Names: GTR

SUMMARY:
This randomized, controlled split-mouth study will include 24-40 patients. After GTR, a test and a control side will be selected by means of a computer-generated randomization list. Test sides will receive a periodontal dressing (Coepak") for 14 days and the control sides will receive no periodontal dressing. After 14 days the periodontal dressing will be removed and the pain experience will be recorded. After 6-9 months, the clinical periodontal parameters will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.

  * A minimum of 18 teeth, wisdom teeth excluded.
  * Previously untreated moderate chronic periodontitis (Armitage 1999) with radiographic evidence of generalized alveolar bone loss >30%.
  * Presence of at least one pocket with probing pocket depth (PPD) ≥6 mm per quadrant, which was BOP.
  * Presence of at least three teeth per quadrant.

Exclusion Criteria:

* Periodontal treatment in the last 3 years.

  * Antibiotic intake 6 months before • the screening visit.
  * Pregnancy. Systemic diseases with an impact on periodontal healing (e.g. Dia- betes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Pain experience | 14 days
  pain experience will be measured 14 days after GTR procedure; when the dressing is removed. Participants have to fill a VAS score out about pain intensity on a scale from 0 to 10 (0 = no pain, 5 = moderate pain and 10 = worst imaginable pain) and the amount of pain medication taken will be recorded

SECONDARY OUTCOMES:
Probing pocket depth | 6 months
  changes in periodontal probing pocket depth in mm
Attachment level | 6 months
  changes in clinical attachment level in mm

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abu-Ta'a, Principal Investigator — Department of Dental sciences, Faculty of Graduate Studies, Arab American University (AAUP)
Locations (1):
- Mahmoud Abu-Ta'a, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided